CLINICAL TRIAL: NCT06485102
Title: Differences of the Postoperative Outcome for Carotid Surgery Patients Treated by Either Male or Female Surgeons
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Augsburg (Other)
Collaborators: Epidemiology, Faculty of Medicine, University of Augsburg (Unknown)
Responsible Party: Sponsor
Other Study IDs: CAROTIS
Record Dates: First submitted 2024-01-29; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Carotid Stenosis
Keywords: Carotid Artery; Apoplexy; Surgical outcome; Gender specific outcome; Surgeon gender
MeSH Terms: conditions — Carotid Stenosis; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing surgery: A retrospective data collection will be conducted for all the patients, that between jan. 2012 and dec. 2023, were operated because of a carotid stenosis in the University Clinic for Vascular and Endovascular Surgery in Augsburg. This stenosis may have been symptomatic or asymptomatic. The surgery must respect the latest quality assurance for that period.
  Interventions: Procedure: Carotid Surgery in patients with symptomatic or asymptomatic stenosis

INTERVENTIONS:
Procedure: Carotid Surgery in patients with symptomatic or asymptomatic stenosis — Carotid Surgery in patients with symptomatic or asymptomatic stenosis

SUMMARY:
This research will focus on the differences of the postoperative outcome for carotid surgery patients treated by either male or female surgeons. Since 2012, in Germany, the surgical treatment of carotid stenosis has an established quality assurance, making the thematic especially suitable for testing the surgical results of either male or female surgeons.

DETAILED DESCRIPTION:
Data about physician gender having impact on the treatment quality of a patient first appeared in 1999, the publication being about patients with breast cancer. This discussion was resumed in 2016 when Y. Tsugawa et. al showed that female doctors have, in comparison to male doctors, better treatment results. Primary outcomes for the study were mortality and readmissions, which were lower if the treatment has been done by a female doctor. Until today, there are only a few reports about the role of physician gender, especially that of surgeons, in the treatment quality. Studies like the ones from Blohm et. al and Wallis et. al show that female surgeons have a better outcome and a lower mortality, 30 days after the surgery. Wallis et. al also showed that the correlation between male surgeons and female patients have the worst results].

None of the studies that were written until today focussed on carotid surgery. Since 2012, in Germany, the surgical treatment of carotid stenosis has an established quality assurance, with specific documentation and a standard surgical course of action. This is why we consider that this surgery is especially suitable for comparison of results, depending on surgeon genders.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 years
* All the patients that had a carotid revascularisation between jan. 2012 and dec. 2023.

Exclusion Criteria:

- No quality assurance

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — The impact of surgeons' gender on the postoperative outcomes. The impact of surgeons' team gender on the postoperative outcome. The connection between patients' gender and surgeons' gender regarding postoperative outcome.
Study Population: A retrospective data collection will be conducted for all the patients, that between jan. 2012 and dec. 2023, were operated because of a carotid stenosis in the University Clinic for Vascular and Endovascular Surgery in Augsburg. This stenosis may have been symptomatic or asymptomatic. The surgery must respect the latest quality assurance for that period.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The impact of surgeons' gender, team gender and patients gender on postoperative apoplexy | 0-30 days
  stroke [observed in a time frame of 30 days after the operation]
The impact of surgeons' gender team gender and patients gender on postoperative peripheral nerve lesions | 0-30 days
  Impairment of peripheral cervial nerves [observed in a time frame of 30 days after the operation]
The impact of surgeons' gender team gender and patients gender on reinterventions | 0-30 days
  Number of patients with surgical revision
The impact of surgeons' gender team gender and patients gender on procedure related death | 0-30 days
  Number of patients who died following surgery

SECONDARY OUTCOMES:
The impact of surgeons' gender team gender and patients gender on procedure time | 0-30 days
  Duration of surgery measured in minutes
The impact of surgeons' gender team gender and patients gender on the length of stay | 0-30 days
  length of stay in days

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Hyhlik-Duerr, Prof., Study Chair — University Hospital Augsburg Vascular Surgery
Locations (1):
- University Hospital Augsburg, Augsburg, Germany

IPD SHARING:
Plan to Share IPD: No
anonymous study design